CLINICAL TRIAL: NCT00676832
Title: A Multi-Center, Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging Study of COLAL-PRED in the Treatment of Patients With Moderate to Severe Ulcerative Colitis
Brief Title: Study of COLAL-PRED to Treat Moderate to Severe Ulcerative Colitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Prometheus Laboratories (Industry)
Responsible Party: Emil Chuang, Sr. Medical Director, GI Clinical Dev & Med Affairs, Prometheus Laboratories, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 08CP01
Record Dates: First submitted 2008-05-09; First posted 2008-05-13 (Estimated); Last update posted 2010-09-29 (Estimated); Status verified 2010-09

CONDITIONS: Colitis, Ulcerative
Keywords: colitis; ulcerative; moderate; severe
MeSH Terms: conditions — Colitis, Ulcerative; Colitis; Ulcer; Lymphoma, Follicular | interventions — Methylprednisolone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Group 1 (Placebo Comparator)
  Interventions: Drug: Placebo
- Group 2 (Experimental)
  Interventions: Drug: COLAL-PRED
- Group 3 (Experimental)
  Interventions: Drug: COLAL-PRED
- Group 4 (Experimental)
  Interventions: Drug: COLAL-PRED
- Group 5 (Experimental)
  Interventions: Drug: COLAL-PRED

INTERVENTIONS:
Drug: Placebo — Placebo solid capsule dosage form administered orally once daily.
  Other Names: prednisolone sodium metasulfobenzoate (PMSBS)
  Arms: Group 1
Drug: COLAL-PRED — The study is a double-blinded and results have not been unblinded. Patients were randomized to one of four doses. A solid capsule dosage form was administered orally once daily at doses of 40 mg, 60 mg, 80 mg, or 120 mg.
  Other Names: prednisolone sodium metasulfobenzoate (PMSBS)
  Arms: Group 2; Group 3; Group 4; Group 5

SUMMARY:
The purpose of this study is to determine whether COLAL-PRED is a safe and effective treatment for patients with moderate to severe ulcerative colitis.

DETAILED DESCRIPTION:
This is a multi-center, randomized, double-blind, placebo-controlled, parallel-design, dose-ranging study. Eligible patients with a DAI score of 6 to 10 (inclusive), plus endoscopic evidence of moderate to severe ulcerative colitis as assessed by flexible sigmoidoscopy, unless colonoscopy is clinically indicated, and rectal bleeding will be randomized to placebo or one of four doses of COLAL-PRED (equivalent to 40, 60, 80, or 120 mg of prednisolone). The effectiveness and safety of COLAL-PRED will be evaluated at baseline, and after 2 weeks and 4 weeks of treatment. Additional follow-up measurements will take place 7 days post cessation of treatment.

The systemic absorption of COLAL-PRED will be determined by measuring blood levels of prednisolone, prednisolone sodium metasulfobenzoate (PMSBS) and metasulfobenzoate at Week 4.

Hypothalamic-pituitary-adrenocortical (HPA) axis response will be monitored by measuring morning serum cortisol levels at Baseline, Week 2, Week 4, and at follow-up visit and cortisol levels following adrenocorticotrophic hormone (ACTH) stimulation testing at Baseline and Week 4.

ELIGIBILITY:
Inclusion Criteria:

* Females must be of non-childbearing potential evidenced by being surgically sterile, postmenopausal for at least 12 months or be using acceptable contraception methods such as contraceptive pill, or two forms of barrier contraception.
* Disease Activity Index (DAI) Score of 6-10 (inclusive) at the Baseline Visit.
* Previous colonoscopic and biopsy diagnosis of ulcerative colitis with negative evaluation of the ileum within 3 years of the screening visit.
* Endoscopic evidence of moderate or severe mucosal disease as assessed by flexible sigmoidoscopy, with a minimum confirmed diagnosis of moderate ulcerative colitis.
* The following concomitant prescription medications for ulcerative colitis are permitted if the following conditions are met:

  1. Oral 5-aminosalicylic acid (5-ASA )therapy if the following 2 criteria are met:

     1. Must be on a stable dose 2 weeks prior to baseline
     2. Must maintain the stable dose until treatment end.
  2. Azathioprine or 6-mercaptopurine or methotrexate if the 4 following criteria are met:

     1. On therapy continually for at least 3 months prior to baseline.
     2. And on a stable dose for at least 2 weeks prior to baseline.
     3. And must maintain the stable dose until the end of study drug treatment.

Exclusion Criteria:

* History of colonic or rectal surgery, excluding hemorrhoidal surgery or an appendectomy.
* Pregnant or breast-feeding females.
* Diagnosis of diabetes, heart failure, unstable angina, hepatic cirrhosis, kidney failure, adrenocortical insufficiency, or any other unstable medical condition.
* Known hypersensitivity to corticosteroids
* Use of oral 5-aminosalicylic acid (5-ASA) or oral corticosteroids during the immediate screening period.
* Use of immunosuppressive drugs or antibiotics at any time within four weeks prior to screening.
* Diagnosis of Crohn's disease; indeterminate colitis; microscopic colitis; ischemic, infectious (e.g., salmonella, shigella, etc.), or amebic colitis; or gonococcal proctitis; Clostridium difficile colitis.
* History of tuberculosis or HIV
* Clinically significant abnormal laboratory test results, unless regarded by the Investigator as related to ulcerative colitis
* History of alcohol or drug abuse
* Known malignancy or history of malignancy that would reduce life expectancy
* Recent immunization with live viral vaccines
* History of or active peptic ulcer disease or gastritis
* Generalized infections such as systemic fungal or hepatitis B or C
* History of steroid induced severe hypertension, steroid-induced psychosis, or any other severe steroid-related adverse reaction

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2008-05; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
The proportion of patients with Complete Response at Week 4 defined as a decrease from baseline in the DAI score by ≥ 30% or ≥ 3 points, and with a decrease in the rectal bleeding subscore of ≥ 1 or an absolute rectal bleeding sub-score of 0 or 1. | Week 4 of the study or at time of withdrawal

SECONDARY OUTCOMES:
The proportion of patients in Clinical Remission defined as a DAI score of ≤ 2 points, with no-individual DAI sub-score > 1 at Week 4. Patients in remission by this definition will have a rectal bleeding DAI sub-score of either 0 or 1. | Week 4

CONTACTS AND LOCATIONS:
Overall Officials: David T. Rubin, M.D., Principal Investigator — The University of Chicago Hospitals
Locations (89):
- United States (89):
  - Prometheus Investigational Site #059, Birmingham, Alabama
  - Prometheus Investigational Site #042, Huntsville, Alabama
  - Prometheus Investigational Site #081, Huntsville, Alabama
  - Prometheus Investigational Site #033, Montgomery, Alabama
  - Prometheus Investigational Site #067, Scottsdale, Arizona
  - Prometheus Investigational Site #090, Tucson, Arizona
  - Prometheus Investigational Site #068, Jonesboro, Arkansas
  - Prometheus Investigational Site #065, Little Rock, Arkansas
  - Prometheus Investigational Site #093, Lowell, Arkansas
  - Prometheus Investigational Site 062, Fresno, California
  - Prometheus Investigational Site #057, Madera, California
  - Prometheus Investigational Site #060, Palm Springs, California
  - Prometheus Investigational Site #095, Roseville, California
  - Prometheus Investigational Site #003, San Carlos, California
  - Prometheus Investigational Site #022, San Diego, California
  - Prometheus Investigational Site #052, Santa Monica, California
  - Prometheus Investigational Site #086, West Covina, California
  - Prometheus Investigational Site #097, Lafayette, Colorado
  - Prometheus Investigational Site #006, Littleton, Colorado
  - Prometheus Investigational SIte #036, Thornton, Colorado
  - Prometheus Investigational Site #031, Hamden, Connecticut
  - Prometheus Investigational Site #083, Hartford, Connecticut
  - Prometheus Investigational Site #023, Cape Coral, Florida
  - Prometheus Investigational Site #075, Cape Coral, Florida
  - Prometheus Investigational Site #076, Hollywood, Florida
  - Prometheus Investigational Site #007, Jacksonville, Florida
  - Prometheus Investigational Site #008, Miami, Florida
  - Prometheus Investigational Site #027, Sarasota, Florida
  - Prometheus Investigational Site #066, Winter Park, Florida
  - Prometheus Investigational Site #005, Atlanta, Georgia
  - Prometheus Investigational Site #044, Atlanta, Georgia
  - Prometheus Investigational Site #010, Arlington Heights, Illinois
  - Prometheus Investigational Site 041, Chicago, Illinois
  - Prometheus Investigational Site # 001, Chicago, Illinois
  - Prometheus Investigational Site #089, Peoria, Illinois
  - Prometheus Investigational Site #059, Anderson, Indiana
  - Prometheus Investigational Site #015, Davenport, Iowa
  - Prometheus Investigational Site #051, Topeka, Kansas
  - Prometheus Investigational Site #039, Baton Rouge, Louisiana
  - Prometheus Investigational Site #061, Lafayette, Louisiana
  - Prometheus Investigational Site 092, New Orleans, Louisiana
  - Prometheus Investigational Site 100, Shreveport, Louisiana
  - Prometheus Investigational Site #016, Chevy Chase, Maryland
  - Prometheus Investigational Site #046, Hagerstown, Maryland
  - Prometheus Investigational Site #035, Laurel, Maryland
  - Prometheus Investigational Site #025, Lutherville, Maryland
  - Prometheus Investigational Site #037, Boston, Massachusetts
  - Prometheus Investigational Site #018, Braintree, Massachusetts
  - Prometheus Investigational Site #091, Southbridge, Massachusetts
  - Prometheus Investigational Site # 050, Chesterfield, Michigan
  - Prometheus Investigational Site #011, Novi, Michigan
  - Prometheus Investigational Site #072, Wyoming, Michigan
  - Prometheus Investigational Site #098, Plymouth, Minnesota
  - Prometheus Investigational Site #021, Jackson, Mississippi
  - Prometheus Investigational Site #019, Mexico, Missouri
  - Prometheus Investigational Site #017, Lebanon, New Hampshire
  - Prometheus Investigational Site #014, Cedar Knolls, New Jersey
  - Prometheus Investigational Site #009, Egg Harbor, New Jersey
  - Prometheus Investigational Site #063, Ocean City, New Jersey
  - Prometheus Investigational Site #080, Brooklyn, New York
  - Prometheus Investigational Site #002, Great Neck, New York
  - Prometheus Investigational Site #079, Rochester, New York
  - Prometheus Investigational Site 043, Rockville Centre, New York
  - Prometheus Investigational Site 087, Stony Brook, New York
  - Prometheus Investigational Site #013, Charlotte, North Carolina
  - Prometheus Investigational Site #047, Greenville, North Carolina
  - Prometheus Investigational Site #058, Wilmington, North Carolina
  - Prometheus Investigational Site #069, Columbus, Ohio
  - Prometheus Investigational Site #070, Dayton, Ohio
  - Prometheus Investigational Site #064, Dayton, Ohio
  - Prometheus Investigational Site #055, Mentor, Ohio
  - Prometheus Investigational Site #094, Westlake, Ohio
  - Prometheus Investigational Site #028, Tulsa, Oklahoma
  - Prometheus Investigational Site #049, Tulsa, Oklahoma
  - Prometheus Investigational Site #030, Philadelphia, Pennsylvania
  - Prometheus Investigational Site #038, Philadelphia, Pennsylvania
  - Prometheus Investigational Site #034, Sayre, Pennsylvania
  - Prometheus Investigational Site #045, Charleston, South Carolina
  - Prometheus Investigational Site #084, Franklin, Tennessee
  - Prometheus Investigational Site #020, Germantown, Tennessee
  - Prometheus Investigational Site #053, Nashville, Tennessee
  - Prometheus Investigational Site #074, Union City, Tennessee
  - Prometheus Investigational Site 101, Denton, Texas
  - Prometheus Investigational Site #071, Plano, Texas
  - Prometheus Investigational Site #026, San Antonio, Texas
  - Prometheus Investigational Site #073, San Antonio, Texas
  - Prometheus Investigational Site #082, Sugar Land, Texas
  - Prometheus Investigational Site #012, Ogden, Utah
  - Prometheus Investigational Site #040, Seattle, Washington